CLINICAL TRIAL: NCT02106871
Title: Phase I Assessment of NO Mediated Signaling in Cancer Cachexia
Brief Title: Study of Sildenafil as a Therapy for Fatigue in Pancreatic Cancer
Acronym: PCC
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study did not get funded. Study never started
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 13-0409
Record Dates: First submitted 2014-01-30; First posted 2014-04-08 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Pancreatic Cancer; Cholangiocarcinoma
Keywords: cancer; pancreas; cholangiocarcinoma; fatigue; sildenafil; lean mass; muscle
MeSH Terms: conditions — Pancreatic Neoplasms; Cholangiocarcinoma; Neoplasms; Fatigue | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo daily for 4 weeks
  Interventions: Drug: Sildenafil
- Sildenafil (Active Comparator): 50mg sildenafil daily for 4 weeks
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Sildenafil — 50mg of Sildenafil daily for 4 weeks
  Other Names: Viagra

SUMMARY:
Investigation of the effects of daily sildenafil on patients with pancreatic or cholangiocarcinoma cancer undergoing treatment.

DETAILED DESCRIPTION:
This is a double-blinded, placebo-controlled trial in men and women, 40-75 years old, diagnosed with pancreatic or cholangiocarcinoma cancer. Patients will receive placebo or sildenafil daily for 4 weeks during their initial chemotherapy cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, aged 40-75 years.
2. Diagnosed with Stage III or IV pancreatic or cholangiocarcinoma receiving the following therapy:

   * Neoadjuvant chemotherapy
   * Surgical resection followed by chemotherapy.
3. Able to comprehend risks and sign a consent form.
4. Performance Status of 0-2.

Exclusion Criteria:

1. Significant renal or heart disease or any acute metabolic disease.
2. Evidence of hepatitis as indicated by a 3-fold increase in of 2 out of 3 liver enzymes.
3. Diabetes mellitus or other untreated endocrine disease.
4. Recent (within 3 months) treatment with anabolic steroids.
5. Ongoing anticoagulant therapy.
6. Androgen secreting tumors of the ovary and adrenal or any ovarian tumor (e.g., Sertoli-Leydig).
7. Polycystic ovary syndrome (PCOS) and/or hyperthecosis.
8. Non-classical adrenal hyperplasia.
9. Cushing's syndrome.
10. Glucocorticoid resistance.
11. Pregnancy.
12. Hyperprolactinoma, hypothyroidism.
13. Use of nitrates.
14. Use of alpha blockers.
15. Use of protease inhibitors.
16. Use of cytochrome p450 inhibitors.
17. Systolic blood pressure <100 or >150, diastolic blood pressure <60 or >90. This range is smaller than the acceptable range stated in the prescribing information for sildenafil (>90/50 and <170/110).
18. Peripheral vascular disease.
19. Use of a phosphodiesterase 5 inhibitor.
20. Any other circumstance deemed exclusionary by the PI or study physician.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Lean Body Mass | 4 weeks
  Lean body mass will be measured by DEXA scan
Skeletal Muscle Fatigue | 4 weeks
  Skeletal muscle fatigue will be measured by leg dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Melinda Sheffield-Moore, PhD, Principal Investigator — University of Texas
Locations (1):
- The University of Texas Medical Branch, Galveston, Texas, United States